CLINICAL TRIAL: NCT06106100
Title: Efficacy and Safety of Endoscopic Anti-reflux Mucosal Ablation Therapy for Gastroesophageal Reflux Disease: a Single Blind Randomized Sham Controlled Trial
Brief Title: Anti-reflux Mucosal Ablation Therapy Randomized Sham Control Trial for Gastroesophageal Reflux Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112122-F
Record Dates: First submitted 2023-10-22; First posted 2023-10-30 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-09

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antireflux mucosal ablation (Active Comparator): In patients fulfilling the inclusion criteria and being randomized for ARMA, retroflexion endoscopy to visualize the cardia is performed, followed by mucosa markings with straight-fire APC catheter (ERBE Electromedizin, Tübingen, Germany) in forced coagulation mode (VIO300D, ERBE Electromedizin, Tübingen, Germany, 20W). The marking site at 1-cm and 2-cm distal to squamocolumnar junction at anterior-posterior and lesser curvature site, respectively, sparing the greater curvature site of cardia, is done. After marking, mucosal ablation (forced coagulation mode, 1L/min, 80W) is performed at marking site in a hoarse-shoe shape. Adequate ablation depth is defined as reaching the submucosal layer with blackish discolored tissue with carbonization
  Interventions: Procedure: Antireflux mucosal ablation
- Sham procedure (Sham Comparator): In patients fulfilling the inclusion criteria and being randomized for sham procedure, retroflexion endoscopy to visualize the cardia is performed. Using the straight-fire APC catheter to touch the marking sites similar to the treatment group without electrocauterization is performed
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Antireflux mucosal ablation — Patients are instructed to fast for 6 hours pre-procedurally, which are performed under intravenous propofol sedation. Retroflexion endoscopy to visualize the cardia is performed, followed by mucosa markings with straight-fire APC catheter (ERBE Electromedizin, Tübingen, Germany) in forced coagulation mode (VIO300D, ERBE Electromedizin, Tübingen, Germany, 20W). The marking site at 1-cm and 2-cm distal to squamocolumnar junction at anterior-posterior and lesser curvature site, respectively, sparing the greater curvature site of cardia, is done. After marking, mucosal ablation (forced coagulation mode, 1L/min, 80W) is performed at marking site in a hoarse-shoe shape. Adequate ablation depth is defined as reaching the submucosal layer with blackish discolored tissue with carbonization
  Arms: Antireflux mucosal ablation
Procedure: Sham procedure — Patients are instructed to fast for 6 hours pre-procedurally, which are performed under intravenous propofol sedation. Retroflexion endoscopy to visualize the cardia is performed. Using the straight-fire APC catheter to touch the marking sites similar to the treatment group without electrocauterization is performed.
  Arms: Sham procedure

SUMMARY:
The goal of this randomized clinical trial is to investigate the efficacy and safety of antireflux mucosal ablation (ARMA) for patients with refractory gastroesophageal reflux disease (GERD). The trial aim to evaluate :

* Efficacy of ARMA comparing with medical treatment alone (proton pump inhibitor (PPI)), using GERD-Health Related Quality of Life Questionnaire (GERD- HRQL questionnaire), improvement of acid exposure time and DeMeester score
* Safety and complications of ARMA Participants will be randomly divided into 2 groups. The intervention group will be undergone ARMA, and the control group will be undergone sham endoscopic treatment.

The primary endpoint will be symptoms relief (GERD-HRQL decreases > 50%). The secondary endpoint will be dosage adjustment of PPI, complications, improvement of acid exposure time and DeMeester score.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years old
* History of GERD for over 6 months, who had received PPIs for over 6 months but still had symptoms of typical GERD symptoms (GERD-HRQL score of >8, acid reflux sensation or heartburn), and/or other symptoms as lump throat, night cough, acid related chest tightness (without other possible explanation of these symptoms)
* Acid exposure time > 6%
* DeMeester score ≥ 14.72

Exclusion Criteria:

* Pregnancy
* BMI>=35
* Hiatal hernia > 2cm or Flap Valve Hill grade III/IV
* GERD LA grade C/D or esophageal ulcer
* Abnormal anatomy of esophagus (esophagectomy, stricture, diverticulum)
* Barrett's esophagus with dysplasia
* Esophageal motility disorders
* History of gastroparesis
* Cirrhosis
* Esophageal and gastric varices
* Previous gastric surgery and anti-reflux procedures
* History of scleroderma or dermatomyositis
* Coagulation disorders (Bleeding tendency and coagulopathy)
* History of oncological disease (not active within 2 years)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of gastroesophageal reflux disease symptoms | 3 months
  Clinical success is defined as more than 50% improvement of the GERD-HRQL questionnaire at 3 months after the ARMA procedure. The results are from minimal 0 points up to 50 points. The higher the points, the greater the symptoms.

SECONDARY OUTCOMES:
Complication rate | 12 months
  Recording of all complications related to the ARMA procedure
PPI dependency | 12 months
  Requirement and dose of PPI at 3, 6 and 12 months after ARMA
Changes in acid exposure time | 12 months
  Changes in acid exposure time in 24 pH meter at 3 and 12 months after ARMA
Changes in DeMeester score | 12 months
  Changes in DeMeester score in 24 pH meter at 3 and 12 months after ARMA. A DeMeester score of ≤ 14.72 is considered physiological.
Changes in lower esophageal sphincter pressure | 12 months
  Changes in lower esophageal sphincter pressure in high resolution manometry at 3 and 12 months after ARMA